CLINICAL TRIAL: NCT05401123
Title: Comparison of Breast Milk Content in Mothers Using a Expressing Pump and Milking by Hand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, associate oroffesor, Gazi University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: mineis001
Record Dates: First submitted 2022-04-21; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Breastfeeding; Human Milk
Keywords: breast milk; breastfeeding; milk contents; human milk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: breasting pump
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of Breast Milk Content in Mothers Using a Expressing Pump and Milking by Hand (Experimental): Randomization In order to ensure similarity between groups; Stratified block randomization was used to assign the women in the sample group to the experimental and control groups. According to the stratified block randomization method, the imbalances that may occur in the experimental and control groups are limited. In this method, block randomization is performed within each stratum after stratification according to risk factors (Akın & Koçoğlu, 2017; Kanık, Taşdelen & Erdoğan, 2011). Since the mode of delivery affects the content of breast milk, women will be divided into two layers as vaginal delivery and cesarean section in terms of delivery type (Table 1).
  In order to determine the strata group of the woman who was found to meet the research criteria and accepted to participate in the study, a list of assignments was created through the website www.randomizer.org by making 6 blocks with a combination of 4 .
  Experiment: A Control: B
  Interventions: Device: milking pump

INTERVENTIONS:
Device: milking pump — n the study, all mothers who come to the Lactation/Relactation outpatient clinic will be informed about the study, and mothers who accept the study will have to fill out the "Conformity to Criteria Form" created by the researcher. Between the ages of 20-35, postpartum 1-5. Participants who gave birth after the 37th week of pregnancy, did not have literacy problems, mental disabilities and communication problems, did not have chronic diseases, did not use any medication, and volunteered to participate in the study will be included in the study. by milking, 2 ml of first milk will be taken from the participants in the control group (via the milking pump). The collected milk will be taken to the laboratory for analysis by the researcher.

SUMMARY:
The researchers planned this study to compare the effects of breast pumps, which are frequently used today, and manual milking after manual massage on the change in milk content when breast and breastfeeding problems develop.

DETAILED DESCRIPTION:
Comparison of the methods used to solve the milk secretion and breastfeeding problems of the participants in the postpartum period; effective and uncomplicated methods should be put forward. Today, breast milk is expressed by hand using massage or pumps. Both milking techniques used have positive and negative aspects. While there are studies showing that breast milk content is affected by the milking techniques used, there are also studies showing that it does not. This study by the researchers was planned to compare the effects of post-massage pumps and manual milking on the change in milk content. For this reason, it is thought that the researchers will contribute to the literature scientifically and, since it is a doctoral thesis, it can be a guide for future studies on the subject.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 20-35

* Postpartum 1-5. between the day
* Those who gave birth after the 37th week of pregnancy
* The baby does not have any condition that prevents sucking
* Those whose baby is not hospitalized in the neonatal intensive care unit
* Those who do not have literacy problems, mental disabilities and communication problems
* Mothers who agreed to participate in the study voluntarily

Exclusion Criteria:

Those who want to quit working voluntarily

* Inaccessible, cut off communication during operation
* Mothers whose babies were hospitalized during the study
* Hospitalized during the study
* Not completing study post-tests
* Who does not do any milking for a day
* Mothers who express only once a day for two consecutive days

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06-05 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
The protein contents will be analyzed by Miris®️ HMA | 12 week
  Breast milk expressed by hand or by pumping. Milks will defrize, then, will warm and will homogenize using Miris Ultrasonic Processor for 5 seconds, and analyzed for protein content performing Miris®️ HMA. analyzes breast milk content. The results of protein contents will be recorded in the breast milk analysis form.
The ph contents will be analyzed by Miris®️ HMA | 12 week
  Breast milk expressed by hand or by pumping. Milks will defrize, then, will warm and will homogenize using Miris Ultrasonic Processor for 5 seconds, and analyzed for ph content performing Miris®️ HMA. The results of ph contents will be recorded in the breast milk analysis form.
The carbohydrate contents will be analyzed by Miris®️ HMA | 12 week
  Breast milk expressed by hand or by pumping. Milks will defrize, then, will warm and will homogenize using Miris Ultrasonic Processor for 5 seconds, and analyzed for carbohydrate contents, it will be recorded in the breast milk analysis form.

IPD SHARING:
Plan to Share IPD: No